CLINICAL TRIAL: NCT03658187
Title: A Double-blind, Randomized, Placebo-controlled, Cross-over Study to Assess the Acute Effect of IP on hGH Levels in Aging Adults
Brief Title: Assessment of the Acute Effect of IP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DM/171201/HGH
Record Dates: First submitted 2018-08-27; First posted 2018-09-05 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Deficiency Growth Hormone
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 2 tablets orally with water and 2 ml of liquid spray to be kept for 30 sec sublingually, before swallowing. To be taken half an hour before dinner prior to the day of site visit.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: IP
- IP (Experimental): 2 tablets orally with water and 2 ml of liquid spray to be kept for 30 sec sublingually, before swallowing. To be taken half an hour before dinner prior to the day of site visit.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: IP

INTERVENTIONS:
Dietary Supplement: Placebo — Beige-brown powder with speckles in clear enteric coated caplet with berry flavor liquid.
Dietary Supplement: IP — Beige-brown powder with speckles in clear enteric coated caplet with berry flavor liquid.

SUMMARY:
It is a nutraceutical system, consisting of oral tablet and an oral spray called Alpha GPC, which helps your body naturally restore the HGH levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females having age between 40-60 years (both inclusive)
* BMI ≥25 and ≤29.9 kg/m2
* FBS ≤ 120 mg/dl
* Serum hGH levels ≤0.94 ng/ml in females and ≤0.12 in males
* Thyroid Stimulating Hormone ≥ 0.35 and ≤ 5.55 mIU/ml

Exclusion Criteria:

* History of thyroid disorder (Hyper/Hypo).
* Smokers having at least 1 cigarette per day.
* Known hypersensitivity or allergy to one or more of the ingredients of the IP
* Participant suffering from primary or secondary insomnia with/without active treatment.
* Alcoholics as defined by consumption of more than 2 standard alcoholic drinks (more than 30 ml/ day) for past 3 months.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Change in the plasma human growth hormone (hGH) levels in aging individuals | Pre-dose: 0 hours and Post dose: 30, 60, 90,120 mins
  Change in serum hGH levels from baseline

SECONDARY OUTCOMES:
Change on Visual Analogue Score for Fatigue | From Day 0 to Day 1
  Change in Visual Analogue Scale score in IP and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastava, M.D., Study Director — Vedic Lifesciences
Locations (1):
- Vedic Lifesciences Pvt. Ltd, Mumbai, Opp Infinity Mall, India

IPD SHARING:
Plan to Share IPD: No